CLINICAL TRIAL: NCT05219331
Title: Impact of Hydrocephalus Treatment on Persistent Disorder of Consciousness Following Acute Brain Injury
Brief Title: Hydrocephalus Treatment on Persistent Disorder of Consciousness
Acronym: HYCO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RC31/20/0010
Record Dates: First submitted 2022-01-20; First posted 2022-02-02 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Disorder of Consciousness
Keywords: consciousness disorder; hydrocephalus; ventriculoperitoneal shunt; autonomic nervous system
MeSH Terms: conditions — Consciousness Disorders; Hydrocephalus | interventions — Ventriculoperitoneal Shunt

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Disorder of consciousness (Other): Ventriculo peritoneal shunt
  Interventions: Procedure: Ventriculoperitoneal shunt

INTERVENTIONS:
Procedure: Ventriculoperitoneal shunt — Treatment oh hydrocephalus

SUMMARY:
After acute brain injury or haemorrhagic stroke, hydrocephalus might participate to consciousness disorder. We plan to explore whether ventriculoperitoneal shunt insertion improves consciousness in patients with vegetative or minimally conscious state and hydrocephalus. Patients with acute brain injury, persistent consciousness disorder and hydrocephalus will be shunted with a detailed follow-up at 3 months combining: clinical evaluation, FluoroDésoxyGlucose positron emission tomography imaging, high density electroencephalogram, electrocardiogram Holter and sympathetic activity by microneurography.

DETAILED DESCRIPTION:
Persistent disorder of consciousness following acute brain injury is a major public health problem. Advances in intensive care allow a growing number of patients to survive after acute brain injury. However, one third of patients in coma following acute brain injury will not recover a consciousness. To date, no specific treatment has shown its effectiveness in the cognitive recovery of those patients. Few clinical cases suggest that hydrocephalus, which is the impairment of cerebrospinal fluid circulation in the brain, may participate to prolonged disorder of consciousness. Hence treating hydrocephalus with a shunt might improve disorders of consciousness. It is possible to gauge intracranial fluid circulation, that is hydrodynamics quantification, and measure resistance to cerebrospinal fluid outflow. Demonstration of an altered hydrodynamics favours the implantation of a shunt to improve cerebrospinal fluid circulation that might modulate brain region involved in the emergence of consciousness. The study hypothesis is that shunting a patient with persistent disorder of consciousness due to acute brain injury and hydrocephalus might improve his state of consciousness. The neural processes underlying will be assessed through comparative analyses of brain metabolic and electrophysiological signatures.

ELIGIBILITY:
Inclusion Criteria:

* adult, post brain injury persistent disorder of consciousness, hydrocephalus requiring ventriculo-peritoneal shunt.

Exclusion Criteria:

* pregnancy, no consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Coma Recovery Scale-revised scale | 3 months and one years after shunt insertion
  Yield stable estimates of patient consciousness status (higher scores mean better outcome)

SECONDARY OUTCOMES:
18Ffluorodeoxyglucose positron emission tomography | 3 months after shunt insertion
  18Ffluorodeoxyglucose positron emission tomography to measure brain glucose uptake across various brain region involved in consciousness
High density electroencephalogram | 3 months after shunt insertion
  electroencephalogram-based automatic classification to apprehend brain connectivity and conscious states
Holter electrocardiogram and blood pressure | 3 months after shunt insertion
  electrocardiogram recording and analysis and blood pressure to gauge heart rate variability
muscle sympathetic nerve activity | 3 months after shunt insertion
  muscle sympathetic nerve activity measured by microneurography to record the electrical activity of the postganglionic sympathetic nerve from peroneal nerves in the lower limb
catecholamines dosage | 3 months after shunt insertion
  catecholamines dosage in blood

CONTACTS AND LOCATIONS:
Overall Officials: Eric SCHMIDT, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (2):
- France (2):
  - Clinique de Verdaich, Gaillac-Toulza
  - Eric SCHMIDT, Toulouse

IPD SHARING:
Plan to Share IPD: No